CLINICAL TRIAL: NCT06210061
Title: A Comparative Study of Propofol-Fentanyl-Dexmedetomidine and Propofol-Fentanyl-Sevoflurane Anesthesia for Major Spine Surgery Under Somato Sensory- and Motor- Evoked Potential Monitoring
Brief Title: Propofol-Fentanyl-Dexmedetomidine and Propofol-Fentanyl-Sevoflurane Anesthesia for Major Spine Surgery Under Somato Sensory- and Motor- Evoked Potential Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim ElSayed Shahin, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Ain Shams University, Egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FMASU MD206/2023
Record Dates: First submitted 2023-12-23; First posted 2024-01-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Propofol; Fentanyl; Dexmedetomidine; Sevoflurane; Spine Surgery; Somatosensory Evoked Potential; Motor Evoked Potential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Propofol-Fentanyl) (Active Comparator): Anesthesia will be induced with propofol (2mg/kg) and fentanyl (1 ug/kg). Anesthesia will be maintained with propofol and fentanyl infusion, commenced at 10 mg/kg/hr and 0.5 ug/kg/hr respectively and adjusted to keep BIS between 40 & 50 during surgery. Minimal dose of atracurium 0.1 mg/kg will be given at induction to facilitate intubation.
  Interventions: Drug: Propofol-Fentanyl
- Group B (Propofol-Fentanyl-Dexmedetomidine) (Experimental): Anesthesia will be induced with propofol (2mg/kg) and fentanyl (1 ug/kg). Anesthesia will be maintained with propofol and fentanyl infusion, commenced at 10 mg/kg/hr and 0.5 ug/kg/hr respectively and adjusted to keep BIS between 40 & 50 during surgery.
  In addition patients will receive Dexmedetomidine (0.5ug.kg) loading dose infused over 10 mins followed by a constant infusion rate of (0.2ug/kg/hr). Minimal dose of atracurium 0.1 mg/kg will be given at induction to facilitate intubation.
  Interventions: Drug: Propofol-Fentanyl-Dexmedetomidine
- Group C (Propofol-Fentanyl-Sevoflurane) (Experimental): Anesthesia will be induced with propofol (2mg/kg) and fentanyl (1 ug/kg). Anesthesia will be maintained with propofol and fentanyl infusion, commenced at 10 mg/kg/hr and 0.5 ug/kg/hr respectively and adjusted to keep BIS between 40 & 50 during surgery.
  In addition the anesthesia will be maintained with inhalational anesthesia of 50% oxygen , 50% air plus sevoflurane concentration adjusted to keep BIS between 40 & 50 . Minimal dose of atracurium 0.1 mg/kg will be given at induction to facilitate intubation
  Interventions: Drug: Propofol-Fentanyl-Sevoflurane

INTERVENTIONS:
Drug: Propofol-Fentanyl — Anesthesia will be induced with propofol (2mg/kg) and fentanyl (1 ug/kg). Anesthesia will be maintained with propofol and fentanyl infusion, commenced at 10 mg/kg/hr and 0.5 ug/kg/hr respectively and adjusted to keep BIS between 40 & 50 during surgery. Minimal dose of atracurium 0.1 mg/kg will be given at induction to facilitate intubation.
  Arms: Group A (Propofol-Fentanyl)
Drug: Propofol-Fentanyl-Dexmedetomidine — Anesthesia will be induced with propofol (2mg/kg) and fentanyl (1 ug/kg). Anesthesia will be maintained with propofol and fentanyl infusion, commenced at 10 mg/kg/hr and 0.5 ug/kg/hr respectively and adjusted to keep BIS between 40 & 50 during surgery.
  In addition patients will receive Dexmedetomidine (0.5ug.kg) loading dose infused over 10 mins followed by a constant infusion rate of (0.2ug/kg/hr). Minimal dose of atracurium 0.1 mg/kg will be given at induction to facilitate intubation.
  Arms: Group B (Propofol-Fentanyl-Dexmedetomidine)
Drug: Propofol-Fentanyl-Sevoflurane — Anesthesia will be induced with propofol (2mg/kg) and fentanyl (1 ug/kg). Anesthesia will be maintained with propofol and fentanyl infusion, commenced at 10 mg/kg/hr and 0.5 ug/kg/hr respectively and adjusted to keep BIS between 40 & 50 during surgery.
  In addition the anesthesia will be maintained with inhalational anesthesia of 50% oxygen , 50% air plus sevoflurane concentration adjusted to keep BIS between 40 & 50 . Minimal dose of atracurium 0.1 mg/kg will be given at induction to facilitate intubation
  Arms: Group C (Propofol-Fentanyl-Sevoflurane)

SUMMARY:
The objective of this study is to evaluate the effect of adding dexmedetomidine on evoked potentials in adult patients undergoing spinal surgery under intravenous anesthesia

DETAILED DESCRIPTION:
A catastrophic complication of spinal surgery is nerve and spinal cord injury. The incidence of neurological defects after spinal surgery can be reduced from 3.7%-6.9% to less than 1% with proper electrophysiological monitoring.

Somatosensory evoked potentials (SEPs) and motor evoked potentials (MEPs) are currently used as adjunct diagnostic methods in spinal surgery, such as scoliosis surgery and spinal stenosis decompression.

Total intravenous anesthesia (TIVA) with propofol and opioids is commonly used in SEPs and MEPs monitoring as it causes increase in latency in comparison to inhalational anesthetics that cause decrease in amplitude .

The amplitudes of MEPs and SEPs are reduced by halogenated volatile anesthetics, limiting their use in spinal surgery that requires electrophysiological monitoring. When volatile anesthetics did not exceed 0.3MAC, they had little effect on MEPs and SEPs . Martin et al. discovered that volatile agent-based anesthesia has application value during neurophysiological monitoring, such as faster awakening and rapid wake-up tests.

As well, volatile anesthetics can reduce the dosage of propofol. As a result, spinal surgery benefits from combined intravenous inhalation anesthesia. As an adjuvant, dexmedetomidine may be useful in reducing the need for propofol.

Dexmedetomidine is a potent and highly selective alpha-2 agonist. It has the effect of sedation, analgesia, sympatholytic, minimal respiratory depression and possible neuroprotection. Its addition to the anesthetic regimen is believed to have the potential of sparing other hypnotics requirement, especially propofol, thus facilitating MEP and SSEP monitoring while providing the beneficial effects it has.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21-45 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status II and III.
* Undergoing major spine surgery

Exclusion Criteria:

* Refusal of procedure or participation in the study by patients.
* Patients with known history of allergy to one of study drugs
* Patients with nerve conduction pathway injury.
* Severe circulatory or respiratory disease.
* Cognitive or psychiatric illness that leads to inability to cooperate, speak or provide informed consent
* Patients with history of Myasthenia gravis, epilepsy , history of pacemaker implantation .
* Patients who need to be awakened during the procedure.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
The amplitude score of Somato sensory evoked potential | 6 hours postoperatively
  The amplitude score of the waveforms will be measured. More than 50% decrease in the amplitude and more than 10% prolongation of the latency of Compound muscle action potential ( CMAP) from the baseline values will be defined as significant

SECONDARY OUTCOMES:
The latency of Somato sensory evoked potential | 6 hours postoperatively
  The latency of the waveforms will be measured. More than 50% decrease in the amplitude and more than 10% prolongation of the latency of Compound muscle action potential (CMAP) from the baseline values will be defined as significant
The latency of motor evoked potential | 6 hours postoperatively
  The latency of the waveforms will be measured. More than 50% decrease in the amplitude and more than 10% prolongation of the latency of Compound muscle action potential (CMAP) from the baseline values will be defined as significant
The amplitude score of motor evoked potential | 6 hours postoperatively
  The amplitude of the waveforms will be measured. More than 50% decrease in the amplitude and more than 10% prolongation of the latency of Compound muscle action potential (CMAP) from the baseline values will be defined as significant
Intraoperative fentanyl consumption | Intraoperatively
  Fentanyl (1 ug/kg) will be used to induce anesthesia.
Intraoperative propofol consumption | Intraoperatively
  Propofol (2mg/kg) will be used to induce anesthesia
Intraoperative dexmedetomidine consumption | Intraoperatively
  Dexmedetomidine (0.5ug/kg) loading dose infused over 10 mins followed by a constant infusion rate of (0.2ug/kg/hr)
Intraoperative sevoflurane consumption | Intraoperatively
  the anesthesia will be maintained with inhalational anesthesia of 50% oxygen , 50% air plus sevoflurane concentration adjusted to keep BIS between 40 & 50
Changes in heart rate | Till the end of operation
  Heart rate will be assessed immediately before the operation and every 10 minutes in the first 30 minutes of the operation then every 15 minutes till the end of the operation.
Changes in mean arterial pressure | Till the end of operation
  Mean arterial pressure will be assessed immediately before the operation and every 10 minutes in the first 30 minutes of the operation then every 15 minutes till the end of operation
Quality of surgical field | Till the end of operation
  Quality of surgical field will be evaluated every 15 minutes using the surgical field rating (SFR) scale of six points : 5 - massive uncontrollable bleeding, 4 - heavy but controllable bleeding that significantly interfered with dissection, 3 - moderate bleeding that moderately compromised surgical dissection, 2 - moderate bleeding - a nuisance but without interference with accurate dissection, 1 - bleeding, so mild it was not even a surgical nuisance, 0 - no bleeding and virtually bloodless field. Surgical field was graded as good, fair, and poor as: good - SFR scale 0 or 1, fair - SFR scale 2or 3, poor - SFR scale 4 or 5).
Intraoperative bleeding | Intraoperatively
  Intraoperative bleeding will be measured by collecting blood in a marked container of 2500 ml capacity and the blood soaked by gauze pieces [4×4 soaked gauze piece (15 ml blood), completely soaked abdominal towel (150 ml blood)]

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.